CLINICAL TRIAL: NCT01244607
Title: A Proof-of-Principle Study Investigating the Effect of Single Doses of NI-0801 on Nickel Induced Contact Dermatitis
Brief Title: NI-0801 in Allergic Contact Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Allocation: Randomized
Other Study IDs: NI-0801-02
Record Dates: First submitted 2010-11-16; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- NI-0801 (Experimental)
  Interventions: Drug: NI-0801

INTERVENTIONS:
Drug: Placebo — single i.v. administration
  Arms: Placebo
Drug: NI-0801 — single i.v. administration
  Arms: NI-0801

SUMMARY:
The purpose of the study is to assess the effect of a single dose of NI-0801 on the severity of nickel-induced allergic contact dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 and ≤ 70 years
* Either male or a female lacking childbearing potential
* Previously documented nickel allergy

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigator, would interfere with safe completion of the trial or that would prevent subjects from providing informed consent.
* Known or previous diagnosis of malignancy
* Known current active tuberculosis or a history of active TB within 12 months of screening
* Known infection with HIV, Hepatitis B or C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)

PRIMARY OUTCOMES:
Effect of NI-0801 administration on the severity of the cutaneous response to Nickel challenge as measured using the score system of the DKG (Deutsche Kontakt-Allergie Gruppe).

SECONDARY OUTCOMES:
Safety and tolerability of NI-0801 as measured by the incidence and severity of treatment emergent adverse events.